CLINICAL TRIAL: NCT05725317
Title: Clinical Performance Assessment of Two Silicone Hydrogel Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLX679-C001
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Refractive Errors; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LID220365 (OD) / LID006961 (OS) (Other): LID220365 contact lens worn in the right eye (OD), with LID006961 contact lens worn in the left eye (OS), as randomized, for four days. A fresh pair of lenses will be worn each day.
  Interventions: Device: LID220365 contact lens; Device: LID006961 contact lens
- LID006961 (OD) / LID220365 (OS) (Other): LID006961 contact lens worn in the right eye (OD), with LID220365 contact lens worn in the left eye (OS), as randomized, for four days. A fresh pair of lenses will be worn each day.
  Interventions: Device: LID220365 contact lens; Device: LID006961 contact lens

INTERVENTIONS:
Device: LID220365 contact lens — Investigational delefilcon A spherical contact lens made with a modified manufacturing process
Device: LID006961 contact lens — Commercially available delefilcon A spherical contact lens
  Other Names: DAILIES TOTAL1®

SUMMARY:
The purpose of this study is to assess the overall clinical performance of a contact lens made with a modified manufacturing process.

DETAILED DESCRIPTION:
The expected duration of subject participation in the study is approximately 4 days with 2 scheduled visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wearer of spherical soft contact lenses of the same brand in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Manifest cylinder equal to or less than 0.75 diopter (D) in each eye.
* Best corrected visual acuity (BCVA) better than or equal to 0.10 logMAR in each eye.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during study participation.
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Habitual monovision or multifocal contact lens wearers.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (7):
- United States (7):
  - Kindred Optics at Maitland Vision, Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Franklin Park Eye Center PC, Franklin Park, Illinois
  - SUNY College of Optometry Clinical Vision Research Center, New York, New York
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - Optometry Group, PLLC, Memphis, Tennessee
  - Clarke Eyecare Center, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7 investigative sites located in the United States.
Pre-assignment Details: Of the 114 enrolled, 1 participant was exited from the study prior to randomization as a screen failure. This reporting group includes all randomized participants (113).
Units Other Than Participants: eyes
Groups:
- LID220365 (OD) / LID006961 (OS): LID220365 contact lens worn in the right eye (OD), with LID006961 contact lens worn in the left eye (OS), as randomized, for four days. A fresh pair of lenses was worn each day.
- LID006961 (OD) / LID220365 (OS): LID006961 contact lens worn in the right eye (OD), with LID220365 contact lens worn in the left eye (OS), as randomized, for four days. A fresh pair of lenses was worn each day.
Period: Overall Study
Arm/Group | LID220365 (OD) / LID006961 (OS) | LID006961 (OD) / LID220365 (OS)
Started | 56; 112 eyes | 57; 114 eyes
Completed | 56; 112 eyes | 57; 114 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID220365 (OD) / LID006961 (OS) | LID006961 (OD) / LID220365 (OS) | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.2) | 33.8 (7.9) | 33.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 18 | 19 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 46 | 93
  Black or African American | 2 | 4 | 6
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 1 | 1
  Multi-racial | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 51 | 48 | 99

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance Visual Acuity (VA) With Study Lenses at Day 4
Description: VA was assessed for each eye individually at a distance of 4 meters with contact lenses in place using a letter chart. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity.
Time Frame: Day 4
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID220365: LID220365 contact lens worn in the right eye (OD) or left eye (OS), as randomized, for four days. A fresh pair of lenses was worn each day.
- LID006961: LID006961 contact lens worn in the right eye (OD) or left eye (OS), as randomized, for four days. A fresh pair of lenses was worn each day.
Arm/Group | LID220365 | LID006961
Number analyzed (Participants) | 113 | 113
Number analyzed (eyes) | 113 | 113
logMAR | -0.13 (0.006) | -0.13 (0.006)
Statistical Analysis 1: Comparison: LID220365 vs LID006961; Test type: Non-Inferiority — Noninferiority in distance visual acuity was declared if the upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; LS Mean Difference = -0.01, 95% CI 1-sided [upper limit 0.00], Standard Error of Mean 0.004 — LSM results based on mixed effects repeated measures model with both fixed (lens, visit, lens-by-visit interaction and sequence) and random (subject) effects. Difference = LID220365 minus LID006961. Sign is retained with the rounded value

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, approximately 4 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting groups.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID220365 Ocular: Events reported in this group occurred while exposed to the LID220365 contact lens.
- LID006961 Ocular: Events reported in this group occurred while exposed to the LID006961 contact lens.
- Overall Non-Ocular: Events reported in this group occurred while exposed to the study contact lenses.
Arm/Group | Pretreatment | LID220365 Ocular | LID006961 Ocular | Overall Non-Ocular
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/113 | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113 | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 0/113 | 0/113 | 0/113 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT05725317/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT05725317/SAP_001.pdf